CLINICAL TRIAL: NCT00142870
Title: Effects of Bupropion on Marijuana Withdrawal Symptoms
Brief Title: Effectiveness of Bupropion in Treating Marijuana Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: David M. Penetar, McLean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-17275-1; R03-17275-1; DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Marijuana Abuse; Substance-Related Disorders
Keywords: marijuana; treatment
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Placebo Comparator)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — 150 mg, twice a day
  Other Names: Zyban

SUMMARY:
A definable and significant withdrawal syndrome occurs upon cessation of chronic, heavy marijuana use. Bupropion (Zyban) is a medication currently used to treat withdrawal symptoms associated with tobacco use. The purpose of this study is to determine if bupropion will help individuals stop using marijuana.

DETAILED DESCRIPTION:
A definable and significant withdrawal syndrome occurs upon cessation of chronic, heavy marijuana use. This syndrome includes alterations in mood, sleep disturbances, and cognitive performance. Many of nicotine's withdrawal symptoms are similar to those observed with marijuana withdrawal. Bupropion has been shown to be effective in treating nicotine addiction.The purpose of this study is to determine if bupropion is effective in treating marijuana dependent individuals. Specifically, this study will determine if bupropion alleviates withdrawal symptoms associated with marijuana abuse.

Participants in this 21-day, double-blind study will be randomly assigned to receive either bupropion or placebo. Treatment with bupropion will occur for one week before stopping marijuana use (quit day). Bupropion will be administered at 150 mg per day for 3 days, followed by 300 mg per day for the remainder of the study. Quit day will occur on Day 8, at which time participants will be required to remain abstinent from marijuana for the duration of the study. Participants will provide daily urine specimens. Changes in vigilance, memory, reaction time, and psychomotor performance as well as withdrawal symptoms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use and dependence
* Marijuana use of at least 5 times in the past 7 days or more than 25 times per month for the 3 years prior to enrollment
* Unsuccessful in a previous attempt to quit marijuana

Exclusion Criteria:

* Axis I disorder
* Any drug abuse or dependence other than marijuana
* Currently taking antipsychotic or antidepressant medication
* Heavy alcohol drinker (more than 20 drinks per week)
* Current nicotine dependence
* History of a seizure disorder
* Current or prior eating disorder (e.g., bulimia or anorexia nervosa)
* Heavy caffeine use (more than 300 mg per day)
* Life threatening or unstable medical illness
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Withdrawal severity | on a daily basis for 14 days

CONTACTS AND LOCATIONS:
Overall Officials: David M Penetar, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Dept. of Psychiatry, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Penetar DM, Looby AR, Ryan ET, Maywalt MA, Lukas SE. Bupropion reduces some of the symptoms of marihuana withdrawal in chronic marihuana users: a pilot study. Subst Abuse. 2012;6:63-71. doi: 10.4137/SART.S9706. Epub 2012 Jun 25. PMID 22879754
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22879754